CLINICAL TRIAL: NCT05605561
Title: The Effect of Digital Storytelling Applied to Children in the Preoperative Period on Anxiety and Negative Emotional Behaviours
Brief Title: The Effect of Digital Storytelling Applied to Children in Preoperative Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Selver METE İZCİ, Phd Candidate, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pamukkale University HSI; 2022SABE007 (Other Grant/Funding Number: Pamukkale University Scientific Research Projects Coordination Unit)
Record Dates: First submitted 2022-10-31; First posted 2022-11-04 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Child; Preoperative Period
Keywords: children; preoperative period; digital storytelling

STUDY DESIGN:
Who Masked: Participant
Masking Description: In this study, study and control groups were determined using the simple randomization method to prevent selection bias. Patients do not know that they are in the experimental and control groups. The data in the study was collected by the researcher. To prevent bias during data collection, the State Anxiety Scale, which could enable patients to self-report, was used. The research was conducted according to the CONSORT 2010 reporting guideline (Schulz et al., 2010). In order to prevent reporting bias, the research data were evaluated by a statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Digital Story) (Experimental): The web-based digital story preparation process will be completed as a 3-5 minute short film by using pictures, videos, voiceovers and various video editing techniques by the researcher trained in storytelling. The digital story will be prepared in an appropriate format, taking into account the cognitive development and period characteristics of school children (7-12 years old).
  Interventions: Other: Digital Story
- Standard Maintenance Group (No Intervention): It is the standard of care given according to the hospital's policies and procedures.

INTERVENTIONS:
Other: Digital Story — It is the standard of care given according to the hospital's policies and procedures.
  Other Names: Standard Maintenance Group
  Arms: Intervention Group (Digital Story)

SUMMARY:
Digital storytelling is the craft and art of exploring different media and software applications to communicate stories in new and powerful ways using digital media. Because new digital tools are inexpensive and widely available, digital storytelling tends to be highly personal and at the same time universal. All in all, it is a very powerful form of communication. Digital storytelling applications include short (three to five minute) films with pictures, video clips, soundtrack and narration; storytelling performances and talks supported by media slideshows or interactive presentations; and web-based applications, including streaming media, podcasts, and blogs.

When looking at the literature, different approaches to using digital storytelling are seen: it is used in the education of health professionals, in academic education, for digital story development and research, and as a therapeutic care intervention.

Studies on the use of digital stories in the field of health have just begun to gain popularity, and it is noteworthy that the studies in the health services literature are not yet at the desired level and prevalence. Healthcare is a unique environment to use digital storytelling intervention as a therapeutic purpose in addition to gaining knowledge in all our activities. Using digital stories; It is thought that it will provide significant benefits to parents/children and health professionals by filling the gap in the literature in order to reduce the negative emotional behaviors and anxiety of children undergoing day surgery in the preoperative period, as an informative intervention that can attract the attention of their children while having fun.

DETAILED DESCRIPTION:
The type of study planned is randomized controlled experimental design. The study group is divided into two as intervention and control groups. The intervention and control groups will be selected by simple random sampling method from among the volunteer participants who meet the inclusion criteria. Power analysis was performed to determine the sample size. It was observed that the effect size obtained in the reference study (Chow et al. 2017) was quite strong (d=0.96). As a result of the power analysis we performed, assuming that a lower level of effect size could be obtained (d=0.8), it was calculated that 80% power could be obtained at the 95% confidence level when at least 52 people (at least 26 people for each group) were included in the study. Considering that there may be data losses, the sample size was planned as 72 people (36 people for each group), taking approximately 30% more than the number of samples calculated as a result of the power analysis.

ELIGIBILITY:
Inclusion Criteria:

Admission to hospital for day surgery Having internet Access Written informed consent from family and volunteers to participate in the study

Exclusion Criteria:

Children with neurological development and learning problems Children with chronic illness who require special medical care No internet Access

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Children's Emotional Manifestation Scale | Day Surgery Day: In the Surgery Waiting Room
  This scale was developed by Li and Lopez (2005) to measure the emotional responses of children during stressful medical procedures.
  Children's Emotional Manifestation Scale was adapted into Turkish by Mete Izci and Çetinkaya (2020). Turkish version of the Children's Emotional Manifestation scale (T-CEMS) was found to be valid and reliable in order to measure the emotional responses of children before stressful medical procedures or in the preoperative period.
Physiological Measurement Form | Day Surgery Day: In the Surgery Waiting Room
  This form consists of children's physiological measurements (pulse, blood pressure and respiration). Physiological measurements will be based on pulse (60-95 beats/minute), blood pressure (100-120/60-75 mmHg) and respiration (14-22 minutes) values, which are considered normal for the 6-12 age group (Hartman and Cheifetz). 2011).
State Anxiety Scale for Children (How Do I Feel Questionnaire) | Preoperative Clinic: 5-7 days before Day Surgery, Day Surgery Day: In the Surgery Waiting Room,At home: 2 weeks postoperatively
  The Children's State Trait Anxiety Inventory was developed by Spielberger in 1973 for 4th and 6th grade children, and its Turkish validity and reliability was established by Özusta (1995) in 615 children aged 9-12 (Özusta 1995).

CONTACTS AND LOCATIONS:
Overall Officials: Bengü ÇETİNKAYA, Phd,Prof., Study Director — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Pamukkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
no.